CLINICAL TRIAL: NCT04244877
Title: Evaluation of the Therapeutic Effect of Rifaximin on Covert Hepatic Encephalopathy With Underlying Small Intestinal Bacterial Overgrowth and Gastrointestinal Dysmotility in Liver Cirrhosis Patients
Brief Title: Rifaximin's Effect on Covert Hepatic Encephalopathy With SIBO and Gastrointestinal Dysmotility
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was unable to recruit participants..
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, RONNIE FASS, Director, Division of Gastroenterology and Hepatology, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-00550
Record Dates: First submitted 2019-12-27; First posted 2020-01-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis, Liver; Minimal Hepatic Encephalopathy; Small Intestinal Bacterial Overgrowth; Gastrointestinal Motility Disorder
MeSH Terms: conditions — Liver Cirrhosis | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rifaximin (Experimental): Rifaximin 550 mg by mouth twice daily for eight weeks.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Drug: Rifaximin tablet
  Other Names: Xifaxan

SUMMARY:
Small Intestinal Bacterial Overgrowth (SIBO) is a common and increasingly recognized disorder in cirrhosis (30% to 73%). One of the most important predisposing factors of SIBO is small bowel dysmotility. Multiple studies have shown that the presence of SIBO is strongly linked to the pathogenesis of Minimal Hepatic Encephalopathy (MHE) also known as Covert Hepatic Encephalopathy (CHE). Consequently, altering and modulating the intestinal microbiota with ammonia-lowering agents and Rifaximin has been the target treatment strategy in CHE. The aim of this study is to determine the therapeutic effect of Rifaximin on patients with CHE and underlying SIBO while assessing the influence of Rifaximin on small bowel motility. In this prospective interventional study, 40 patients with liver cirrhosis will be screened for Covert Hepatic Encephalopathy (CHE) using neuro-psychometric tests. Patients diagnosed with CHE will undergo breath test (BT) for SIBO screening. Afterwards, wireless motility capsule (The SmartPill) will be performed in all patients with a positive BT. Thereafter, the cirrhotic patients diagnosed with CHE and SIBO will receive Rifaximin 550 mg PO twice daily for eight weeks. At the end of treatment, neuro-psychometric tests will be repeated to evaluate the therapeutic effect on CHE. In addition, BT and SmartPill will be repeated at the completion of the Rifaximin treatment period to assess the effect on small bowel motility. All collected clinical parameters at the end of the study will be compared to baseline values.

DETAILED DESCRIPTION:
Small intestinal bacterial overgrowth (SIBO) is a common and an increasingly recognized disorder in liver cirrhosis, correlating with its severity. The prevalence of SIBO, assessed by the quantification of the bacterial density in the small intestinal aspirate, ranges from 30% to 73%. Multiple physiological derangements leading to SIBO appear in cirrhosis from decreased secretion of gastric acid, impaired mucosal immune response to decreased bile acid, and more importantly, intestinal dysmotility. The latter remains the most common predisposing factor in the pathogenesis of bacterial overgrowth. A recent pilot study using a wireless motility capsule (the SmartPill) demonstrated that patients with cirrhosis have significant delays in small bowel transit that is more pronounced in those with more severe liver disease. Altered small bowel motility in cirrhosis has been attributed to autonomic dysfunction, altered levels of circulating neuropeptides and the effects of inflammatory mediators on gut muscle and the enteric nervous system.

Hepatic Encephalopathy (HE) is a spectrum of neuro-cognitive impairment in cirrhosis that range from abnormal neuropsychiatric testing without clinical evidence of disease (Minimal Hepatic Encephalopathy[MHE]) to varying degrees of overt clinical findings: Overt Hepatic Encephalopathy (OHE). MHE is found in 30-84% of patients with liver cirrhosis. The neuro-cognitive deficit noted in MHE could predispose patient to impaired quality of life (QOL) which translates into lower QOL scores, higher risk of falls, driving problems and difficulties maintaining employment. Previous studies have shown that SIBO is prevalent and strongly linked to the pathogenesis of MHE. Consequently, altering and modulating the intestinal microbiota with ammonia-lowering and gut-selective agents has been the target treatment strategy. Multiple prior studies have evaluated Rifaximin efficacy in MHE and have shown improvements across a variety of study clinical end points including neuropsychiatric and QOL tests. However, the precise mechanism of action of Rifaximin in MHE is unclear. The proposed mechanisms by which Rifaximin may lead to improvement of MHE may be beyond the bactericidal/bacteriostatic effect, resulting in changes in bacterial metabolic function/virulence, to an anti-inflammatory and immune-modulatory effect.

The investigators hypothesize that Rifaximin may have an additional effect on small bowel motility that may be independent of its effect on bacterial overgrowth. The effect may not be necessarily through changes in patient's microbiome but rather through a pro-motility mechanism. The investigators intend to test this hypothesis by comparing the motility at baseline in cirrhotic patients with MHE and clinically significant portal hypertension, before and after treatment of SIBO with Rifaximin.

Aims:

1. To determine the therapeutic effect of Rifaximin on patients with CHE and underlying SIBO and as it is related to small bowel motility.
2. To determine the effect of Rifaximin on small bowel motility by using the SmartPill.

Study Design:

This is a prospective and interventional study. It will be conducted at the Gastroenterology and Hepatology outpatient clinics of MetroHealth Medical Center/Case Western Reserve University. Approximately 40 patients with liver cirrhosis will be assessed for eligibility by their hepatologist. Eligible patients will be referred to an expert psychologist for neuro-psychometric testing to confirm CHE. Then the patients with diagnosed with CHE will undergo Glucose Hydrogen Breath Test (BT) for SIBO screening. Subsequently, wireless motility capsule (the SmartPill) for motility testing will be performed in all patients with positive BT. Thereafter, cirrhotic patients diagnosed with both CHE and SIBO will be prescribed Rifaximin 550 mg PO twice daily for eight weeks. At the end of the treatment period, neuro-psychometric tests will be repeated to evaluate the therapeutic effect on CHE. In addition, BT and the SmartPill will be repeated at the completion of the treatment period with Rifaximin in order to assess the effect on small bowel motility.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis patients between 18-89 years of age, without prior transjugular intrahepatic portosystemic shunt (TIPS) placement or prior overt hepatic encephalopathy.
2. Cirrhosis diagnosed on the basis of liver biopsy, liver stiffness measurement (Fibroscan) or radiological study.
3. CHE diagnosis using pre-defined criteria [two of the following should be abnormal as compared to healthy controls: number connection test A/B (NCT-A/B), Digit Symbol Test (DST), or Block Design Test (BDT)] at least 2 months prior to the start of the study (beyond 2 standard deviation of normal). Testing will be carried out by a trained psychologist.

Exclusion Criteria:

1. Known allergy to rifaximin / rifabutin / rifampin.
2. Use of antibiotics within last 6 weeks
3. Use of lactulose / lactitol, probiotics, L-ornithine- L -aspartate, zinc, metronidazole, or neomycin, within last 6 weeks
4. Use of any drug known to affect gastro-intestinal motility within the previous 2 to 4 weeks (such as, Reglan, Erythromycin, or Domeperidone)
5. Use of drugs such as opiates and antidepressants (except stable doses of selective serotonin re-uptake inhibitors)
6. Patients deemed higher risk for capsule retention including a history of esophageal stricture or Zenker's diverticulum, partial or complete bowel obstruction, known ﬁstulas, known large or numerous diverticula and dementia
7. Diseases associated with poor gastrointestinal motility such as uncontrolled diabetes (A1c > 8%), rheumatological disorders (such as scleroderma and mixed connective tissue disorders [MCT])
8. History of gastrointestinal tract or abdominal surgery
9. Spontaneous peritonitis or other severe infections
10. Colonoscopy or enema treatment within 4 weeks
11. Hepatic encephalopathy with clinical signs
12. Inability to complete neuropsychiatric testing due to hearing loss, poor vision, etc.
13. Poorly compliant patients
14. Rifaximin - Pregnancy Category C- There are no adequate and well controlled studies in pregnant women. Rifaximin has been shown to be teratogenic in rats and rabbits at doses that caused maternal toxicity. Female study subjects of childbearing potential must have a negative pregnancy test and agree to use an acceptable method of contraception throughout the study. Participants that are breastfeeding are excluded.
15. Decompensated cirrhosis (i.e., history of variceal bleeding or ascites)
16. Total bilirubin = 2mg/dL or albumin < 3.5g/dL or international normalized ratio (INR) > 1.7
17. Patients with a calculated glomerular filtration rate (GFR) < 60mL/min/1.73m2
18. Patients with severe hepatic impairment (Child-Pugh score > 7)
19. Patients with untreated viral hepatitis
20. No prior episode of overt HE, not on therapy for overt HE, not on any psycho- active medications apart from stable doses of selective serotonin re-uptake inhibitors.
21. No concurrent use of P-glycoprotein inhibitors (e.g., cyclosporine)
22. Current abuse of alcohol or illicit drugs

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Comparing the effects of Rifaximin on patients with covert hepatic encephalopathy (CHE) and SIBO using neuropsychometric test (NST) and glucose hydrogen breath test (BT) after 8 weeks of Rifaximin. | 8 weeks
  The percent of subjects with improvement on Portosystemic Encephalopathy Syndrome test (PSE) after taking Rifaximin for 8 weeks. The percent of subjects who test negative on glucose breath test (BT) after treatment with Rifaximin.

SECONDARY OUTCOMES:
Improvement in small bowel motility in subjects taking Rifaximin | 8 weeks
  The percent of patients with improvement in small bowel motility as measured by the SmartPill after taking Rifaximin for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — Metrohealth Medical Center/Case Western Reserve University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer TM, Schwacha H, Steinbruckner B, Brinkmann FE, Ditzen AK, Kist M, Blum HE. Diagnosis of small intestinal bacterial overgrowth in patients with cirrhosis of the liver: poor performance of the glucose breath hydrogen test. J Hepatol. 2000 Sep;33(3):382-6. doi: 10.1016/s0168-8278(00)80273-1. PMID 11019993
- [Background] Giannelli V, Di Gregorio V, Iebba V, Giusto M, Schippa S, Merli M, Thalheimer U. Microbiota and the gut-liver axis: bacterial translocation, inflammation and infection in cirrhosis. World J Gastroenterol. 2014 Dec 7;20(45):16795-810. doi: 10.3748/wjg.v20.i45.16795. PMID 25492994
- [Background] Quigley EM, Stanton C, Murphy EF. The gut microbiota and the liver. Pathophysiological and clinical implications. J Hepatol. 2013 May;58(5):1020-7. doi: 10.1016/j.jhep.2012.11.023. Epub 2012 Nov 23. No abstract available. PMID 23183530
- [Background] Thalheimer U, De Iorio F, Capra F, del Mar Lleo M, Zuliani V, Ghidini V, Tafi MC, Caburlotto G, Gennari M, Burroughs AK, Vantini I. Altered intestinal function precedes the appearance of bacterial DNA in serum and ascites in patients with cirrhosis: a pilot study. Eur J Gastroenterol Hepatol. 2010 Oct;22(10):1228-34. doi: 10.1097/MEG.0b013e32833b4b03. PMID 20512041
- [Background] Kakiyama G, Pandak WM, Gillevet PM, Hylemon PB, Heuman DM, Daita K, Takei H, Muto A, Nittono H, Ridlon JM, White MB, Noble NA, Monteith P, Fuchs M, Thacker LR, Sikaroodi M, Bajaj JS. Modulation of the fecal bile acid profile by gut microbiota in cirrhosis. J Hepatol. 2013 May;58(5):949-55. doi: 10.1016/j.jhep.2013.01.003. Epub 2013 Jan 16. PMID 23333527
- [Background] Chander Roland B, Garcia-Tsao G, Ciarleglio MM, Deng Y, Sheth A. Decompensated cirrhotics have slower intestinal transit times as compared with compensated cirrhotics and healthy controls. J Clin Gastroenterol. 2013 Nov-Dec;47(10):888-93. doi: 10.1097/MCG.0b013e31829006bb. PMID 23632359
- [Background] Maheshwari A, Thuluvath PJ. Autonomic neuropathy may be associated with delayed orocaecal transit time in patients with cirrhosis. Auton Neurosci. 2005 Mar 31;118(1-2):135-9. doi: 10.1016/j.autneu.2005.02.003. PMID 15795187
- [Background] Fein BI, Holt PR. Hepatobiliary complications of total parenteral nutrition. J Clin Gastroenterol. 1994 Jan;18(1):62-6. doi: 10.1097/00004836-199401000-00015. PMID 8113589
- [Background] Groeneweg M, Quero JC, De Bruijn I, Hartmann IJ, Essink-bot ML, Hop WC, Schalm SW. Subclinical hepatic encephalopathy impairs daily functioning. Hepatology. 1998 Jul;28(1):45-9. doi: 10.1002/hep.510280108. PMID 9657095
- [Background] Shawcross DL, Wright G, Olde Damink SW, Jalan R. Role of ammonia and inflammation in minimal hepatic encephalopathy. Metab Brain Dis. 2007 Mar;22(1):125-38. doi: 10.1007/s11011-006-9042-1. PMID 17260161
- [Background] Randolph C, Hilsabeck R, Kato A, Kharbanda P, Li YY, Mapelli D, Ravdin LD, Romero-Gomez M, Stracciari A, Weissenborn K; International Society for Hepatic Encephalopathy and Nitrogen Metabolism (ISHEN). Neuropsychological assessment of hepatic encephalopathy: ISHEN practice guidelines. Liver Int. 2009 May;29(5):629-35. doi: 10.1111/j.1478-3231.2009.02009.x. Epub 2009 Mar 19. PMID 19302444
- [Background] Simren M, Stotzer PO. Use and abuse of hydrogen breath tests. Gut. 2006 Mar;55(3):297-303. doi: 10.1136/gut.2005.075127. PMID 16474100
- [Background] Saad RJ, Hasler WL. A technical review and clinical assessment of the wireless motility capsule. Gastroenterol Hepatol (N Y). 2011 Dec;7(12):795-804. PMID 22347818
- [Result] Pande C, Kumar A, Sarin SK. Small-intestinal bacterial overgrowth in cirrhosis is related to the severity of liver disease. Aliment Pharmacol Ther. 2009 Jun 15;29(12):1273-81. doi: 10.1111/j.1365-2036.2009.03994.x. Epub 2009 Mar 6. PMID 19302262
- [Result] Zhang Y, Feng Y, Cao B, Tian Q. Effects of SIBO and rifaximin therapy on MHE caused by hepatic cirrhosis. Int J Clin Exp Med. 2015 Feb 15;8(2):2954-7. eCollection 2015. PMID 25932262
- [Result] Gupta A, Dhiman RK, Kumari S, Rana S, Agarwal R, Duseja A, Chawla Y. Role of small intestinal bacterial overgrowth and delayed gastrointestinal transit time in cirrhotic patients with minimal hepatic encephalopathy. J Hepatol. 2010 Nov;53(5):849-55. doi: 10.1016/j.jhep.2010.05.017. Epub 2010 Jul 17. PMID 20675008
- [Result] Sidhu SS, Goyal O, Mishra BP, Sood A, Chhina RS, Soni RK. Rifaximin improves psychometric performance and health-related quality of life in patients with minimal hepatic encephalopathy (the RIME Trial). Am J Gastroenterol. 2011 Feb;106(2):307-16. doi: 10.1038/ajg.2010.455. Epub 2010 Dec 14. PMID 21157444
- [Result] Bajaj JS, Heuman DM, Wade JB, Gibson DP, Saeian K, Wegelin JA, Hafeezullah M, Bell DE, Sterling RK, Stravitz RT, Fuchs M, Luketic V, Sanyal AJ. Rifaximin improves driving simulator performance in a randomized trial of patients with minimal hepatic encephalopathy. Gastroenterology. 2011 Feb;140(2):478-487.e1. doi: 10.1053/j.gastro.2010.08.061. Epub 2010 Sep 21. PMID 20849805
- [Result] Allampati S, Duarte-Rojo A, Thacker LR, Patidar KR, White MB, Klair JS, John B, Heuman DM, Wade JB, Flud C, O'Shea R, Gavis EA, Unser AB, Bajaj JS. Diagnosis of Minimal Hepatic Encephalopathy Using Stroop EncephalApp: A Multicenter US-Based, Norm-Based Study. Am J Gastroenterol. 2016 Jan;111(1):78-86. doi: 10.1038/ajg.2015.377. Epub 2015 Dec 8. PMID 26644276